CLINICAL TRIAL: NCT03350724
Title: Randomized Controlled Clinical Trial Pilot Study: Patient Outcomes and Gingival Blood Flow Using Laser Doppler Flowmetry Following the Use of Episil on Free Gingival Graft Donor Sites
Brief Title: Patient Outcomes and Gingival Blood Flow Using Laser Doppler Flowmetry Following the Use of Episil on Free Gingival Graft Donor Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jennifer James, Clinical Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-15-0658
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Results first posted 2018-03-20 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Pain From Free Gingival Graft

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- episil wound dressing (Experimental): Episil is a wound dressing material intended for the management of pain and relief of pain by adhering to the mucosal surface of the mouth, soothing oral lesions of various etiologies. episil is an oromucosal liquid that transforms in situ to a bioadhesive oromucosal gel by uptake of small amounts of aqueous fluid.
  Interventions: Device: episil wound dressing
- PeriAcryl90 wound dressing (Active Comparator): PeriAcryl90 is a cyanoacrylate wound dressing.
  Interventions: Device: PeriAcryl90 wound dressing

INTERVENTIONS:
Device: episil wound dressing — Episil is a wound dressing material intended for the management of pain and relief of pain by adhering to the mucosal surface of the mouth, soothing oral lesions of various etiologies. episil is an oromucosal liquid that transforms in situ to a bioadhesive oromucosal gel by uptake of small amounts of aqueous fluid.
  Arms: episil wound dressing
Device: PeriAcryl90 wound dressing — PeriAcryl90 is a cyanoacrylate wound dressing.
  Arms: PeriAcryl90 wound dressing

SUMMARY:
The hypothesis for the present study is that patient-based outcomes and gingival blood flow will be more favorable for the free gingival graft (FGG) donor sites being covered by the test wound dressing material episil compared to the control dressing.

ELIGIBILITY:
Inclusion Criteria:

* patient of record at UTHealth School of Dentistry Houston Texas
* signed treatment plan for a FGG
* the ability to provide research informed consent

Exclusion Criteria:

* any allergies to any of the ingredients in episil including allergies to peanuts, soy or peppermint oil
* smokers
* pregnant or breast feeding women
* inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D James, DMD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (17.2) | 47.1 (15.5) | 46.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 8 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: Postoperative pain will be determined by the subjects recording their postoperative pain threshold using a Visual Analog Scale with scores from 1 to 10, with 1 indicating minimal pain and 10 indicating severe pain. If no pain is present, a score of 0 will be given. The levels of postoperative pain will be classified as none to minimum if the score is "0 to 3," moderate for "4 to 6," and severe for "7 to 10." None to minimal pain will mean little or no discomfort; moderate is any pain that bothers the subject and mildly affects normal function; and severe will be considered any pain that will not be tolerated and may even disrupt the subject's daily functions.
Time Frame: 1 day postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 12 | 6
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.039, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

2. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 2 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 13 | 7
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.037, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

3. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 3 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 14 | 8
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.032, Z-Test for Two Population Proportions

4. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 5 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 11 | 8
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.171, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

5. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 7 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 11 | 9
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.484, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

6. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 10 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 13 | 15
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.368, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

7. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 14 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 17 | 16
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.308, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

8. Primary Outcome: Postoperative Pain as Assessed by Number of Participants With a Score of 0-3 (no to Minimal Pain) on a Visual Analog Scale
Description: as for outcome 1
Time Frame: 21 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 17 | 17
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.999, Z-Test for Two Population Proportions — Unadjusted p-value; Unadjusted p-value

9. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: Postoperative pain will be determined by the subjects recording the number of analgesic pills (Ibuprofen 600mg tablets) taken each day.
Time Frame: 1 day postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 2 [1 to 3] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.015, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

10. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: as for outcome 9
Time Frame: 2 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 2 [1 to 3] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

11. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: as for outcome 9
Time Frame: 3 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 2 [1 to 2] | 2 [2 to 4]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.035, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

12. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: as for outcome 9
Time Frame: 5 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 2 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.444, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

13. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: as for outcome 9
Time Frame: 7 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 2 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.765, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

14. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: as for outcome 9
Time Frame: 10 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.941, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

15. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: as for outcome 9
Time Frame: 14 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 0 [0 to 0] | 1 [0 to 1]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.421, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

16. Primary Outcome: Postoperative Pain as Assessed by the Number of Analgesic Pills Taken Each Day
Description: Postoperative pain will be determined by the subjects recording the number of analgesic pills taken each day.
Time Frame: 21 days postoperatively
Measure: Median (Inter-Quartile Range); unit: number of Ibuprofen 600mg tablets
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
number of Ibuprofen 600mg tablets | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney) — Unadjusted p-value; Unadjusted p-value

17. Secondary Outcome: Gingival Blood Flow as Measured Laser Doppler Flometry (LDF)
Description: The laser Doppler flowmetry (LDF) technique to measure the blood perfusion of the free gingival graft (FGG) donor site. The value reported is blood flow at the FGG donor site (operated site) minus blood flow at the contralateral side of the palate (non-operated site). Perfusion Units (PU) are reported, which is blood flow through a given volume or mass of tissue with the unit of measure mL/100g/min.
Time Frame: baseline (on the day of surgery before surgery)
Measure: Mean (Standard Deviation); unit: mL/100g/min
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
mL/100g/min | -34.7 (126.7) | 5.3 (36.0)
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.22, Paired t-Test — Unadjusted p-value; Unadjusted p-value

18. Secondary Outcome: Gingival Blood Flow as Measured Laser Doppler Flowmetry (LDF)
Description: The laser Doppler flowmetry (LDF) technique to measure the blood perfusion of the FGG donor site. The value reported is blood flow at the FGG donor site (operated site) minus blood flow at the contralateral side of the palate (non-operated site). Perfusion Units (PU) are reported, which is blood flow through a given volume or mass of tissue with the unit of measure mL/100g/min.
Time Frame: 3 days postoperatively
Population: One patient was not able to have Day 3 laser Doppler flowmetry (LDF) readings because of a death in the family, and this patient had to travel out of town for several days.
Measure: Mean (Standard Deviation); unit: mL/100g/min
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 16 | 16
mL/100g/min | 42.5 (132.1) | 50.0 (152.3)
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.882, Paired t-Test — Unadjusted p-value; Unadjusted p-value

19. Secondary Outcome: Gingival Blood Flow as Measured Laser Doppler Flowmetry (LDF)
Description: as for outcome 18
Time Frame: 7 days postoperatively
Measure: Mean (Standard Deviation); unit: mL/100g/min
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
mL/100g/min | 203.9 (219.8) | 169.0 (197.7)
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.64, Paired t-Test — Unadjusted p-value; Unadjusted p-value

20. Secondary Outcome: Gingival Blood Flow as Measured Laser Doppler Flowmetry (LDF)
Description: as for outcome 18
Time Frame: 14 days postoperatively
Measure: Mean (Standard Deviation); unit: mL/100g/min
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
mL/100g/min | 266.3 (242.9) | 262.8 (248.1)
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.967, Paired t-Test — Unadjusted p-value; Unadjusted p-value

21. Secondary Outcome: Gingival Blood Flow as Measured Laser Doppler Flowmetry (LDF)
Description: as for outcome 18
Time Frame: 21 days postoperatively
Measure: Mean (Standard Deviation); unit: mL/100g/min
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
mL/100g/min | 151.2 (227.1) | 85.3 (184.7)
Statistical Analysis 1: Comparison: Episil Wound Dressing vs PeriAcryl90 Wound Dressing; Test type: Superiority; p = 0.375, Paired t-Test — Unadjusted p-value; Unadjusted p-value

22. Secondary Outcome: Number of Participants With Re-epithelialization of the FGG Donor Site as Indicated by a Non-invasive Peroxide Test
Description: The non-invasive peroxide test is based on the principle that if the epithelium is discontinuous, the H2O2 diffuses into the connective tissue; the enzyme catalase acts on H2O2 to release water and oxygen: this is clinically shown by the production of bubbles on the wound. 3% H2O2 will be applied to the FGG donor site with a syringe and the appearance of bubbles will be recorded as a dichotomous variable (yes/no).
Time Frame: 3 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 1 | 0

23. Secondary Outcome: Number of Participants With Re-epithelialization of the FGG Donor Site as Indicated by a Non-invasive Peroxide Test
Description: as for outcome 22
Time Frame: 7 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

24. Secondary Outcome: Number of Participants With Re-epithelialization of the FGG Donor Site as Indicated by a Non-invasive Peroxide Test
Description: as for outcome 22
Time Frame: 14 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

25. Secondary Outcome: Number of Participants With Re-epithelialization of the FGG Donor Site as Indicated by a Non-invasive Peroxide Test
Description: as for outcome 22
Time Frame: 21 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
Number analyzed (Participants) | 17 | 17
Participants | 6 | 5

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Episil Wound Dressing | PeriAcryl90 Wound Dressing
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03350724/Prot_SAP_000.pdf